CLINICAL TRIAL: NCT00398996
Title: Study to Compare Three Existing Starting Points of ART Initiation in HIV/TB Co-infected Patients
Brief Title: A Study to Compare Three Existing Starting Points of Anti-Retroviral Therapy (ART) Initiation in HIV/Tuberculosis (TB) Co-infected Patients
Acronym: SAPIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Responsible Party: Director: Prof Salim S Abdool Karim, CAPRISA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPRISA 003
Record Dates: First submitted 2006-11-07; First posted 2006-11-14 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: HIV Infections; Tuberculosis
Keywords: antiretroviral therapy; HIV; Opportunistic infections; CD4; Viral load; TB/HIV co infection; Treatment Naive
MeSH Terms: conditions — HIV Infections; Tuberculosis; Opportunistic Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 - Early integrated-therapy group (Active Comparator): antiretroviral therapy to be initiated within 4 weeks of starting tuberculosis treatment
  Interventions: Drug: Early versus intermediate versus late initiation of ART
- 2 - Late integrated-therapy group (Active Comparator): antiretroviral therapy to be initiated within 4 weeks of completing the intensive phase of tuberculosis treatment
  Interventions: Drug: Early versus intermediate versus late initiation of ART
- 3 - Sequential-therapy group (Active Comparator): Antiretroviral therapy to be initiated within 4 weeks after completing tuberculosis treatment
  Interventions: Drug: Early versus intermediate versus late initiation of ART

INTERVENTIONS:
Drug: Early versus intermediate versus late initiation of ART — Initiation of once daily ddI (400 / 250mg), 3TC (300mg) and EFV (600mg)during the intensive phase of TB therapy or during the continuation phase of TB therapy or once TB therapy has been completed

SUMMARY:
This is a randomized, open-label study comparing three existing treatment strategies of ART initiation in HIV/TB co-infected patients:

Group 1: early initiation of ART with TB treatment, Group 2: initiation of ART upon completion of the intensive phase of TB treatment, Group 3: initiation of ART upon completion of the continuation phase of TB treatment

Approximately 700 men and women ≥ 18 years of age with documented HIV infection and smear-positive pulmonary TB patients will be enrolled. Eligible TB/HIV co-infected patients will be offered antiretroviral therapy (ART), starting at one of the three time points listed above through the CAPRISA AIDS treatment programme which includes extensive counselling and adherence support. The study participants will be followed for 18 months to assess the primary study endpoint of the optimal time to start antiretroviral therapy (ART) in patients on tuberculosis (TB) treatment by comparing clinical status (CD4+ cell count, viral load, opportunistic infections.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients co-infected with TB
* Receiving any one of the standard anti-TB therapy regimens
* All patients must agree to use contraception since they will be on efavirenz.

Exclusion Criteria:

* Entry into the treatment programme is based on a clinical assessment and should patients not be clinically eligible to maintain a treatment regimen,their entry may be deferred or precluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2005-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To measure the incidence of progression to AIDS defining illness or mortality | 18 months

SECONDARY OUTCOMES:
A comparison of CD4+ cell count, viral load, opportunistic infections across the 3 study arms | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Salim S Abdool karim, MBChB, PhD, Principal Investigator — CAPRISA, University of KwaZulu-Natal
Locations (1):
- CAPRISA eThekwini Clinical Research Site, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Background] Abdool-Karim SS, Abdool-Karim Q, Friedland G, Lalloo U, El-Sadr WM; START project. Implementing antiretroviral therapy in resource-constrained settings: opportunities and challenges in integrating HIV and tuberculosis care. AIDS. 2004 Apr 30;18(7):975-9. doi: 10.1097/00002030-200404300-00004. No abstract available. PMID 15096799
- [Result] Abdool Karim SS, Naidoo K, Grobler A, Padayatchi N, Baxter C, Gray A, Gengiah T, Nair G, Bamber S, Singh A, Khan M, Pienaar J, El-Sadr W, Friedland G, Abdool Karim Q. Timing of initiation of antiretroviral drugs during tuberculosis therapy. N Engl J Med. 2010 Feb 25;362(8):697-706. doi: 10.1056/NEJMoa0905848. PMID 20181971
- [Derived] Naidoo K, Yende-Zuma N, Padayatchi N, Naidoo K, Jithoo N, Nair G, Bamber S, Gengiah S, El-Sadr WM, Friedland G, Abdool Karim S. The immune reconstitution inflammatory syndrome after antiretroviral therapy initiation in patients with tuberculosis: findings from the SAPiT trial. Ann Intern Med. 2012 Sep 4;157(5):313-24. doi: 10.7326/0003-4819-157-5-201209040-00004. PMID 22944873
- [Derived] Abdool Karim SS, Naidoo K, Grobler A, Padayatchi N, Baxter C, Gray AL, Gengiah T, Gengiah S, Naidoo A, Jithoo N, Nair G, El-Sadr WM, Friedland G, Abdool Karim Q. Integration of antiretroviral therapy with tuberculosis treatment. N Engl J Med. 2011 Oct 20;365(16):1492-501. doi: 10.1056/NEJMoa1014181. PMID 22010915
- See also: Centre for the AIDS Programme of Research in South Africa's website — http://www.caprisa.org/